CLINICAL TRIAL: NCT07112781
Title: Feasibility Trial of Single-Dose Radiotherapy for Localized Low and Intermediate Risk Prostate Cancer Using Special System of Internal and External Immobilization for Target Motion Mitigation
Brief Title: Feasibility Trial of Single-Dose Radiotherapy for Localized Low and Intermediate Risk Prostate Cancer
Acronym: FAST-ONE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Branch Office of "Hadassah Medical Ltd" (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FAST-ONE
Record Dates: First submitted 2025-08-02; First posted 2025-08-08 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Radiotherapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single-Dose Radiotherapy (SDRT) (Experimental): Patients will be treated using image-guided, volumetric intensity-modulated arc radiotherapy (IGRT-VMAT) with emphasis on normal tissue sparing and delivery accuracy via the use of devices that ensure stability and beam location reproducibility. Patients will be treated with a single fraction at a prescription dose of 24 Gy. In patients in the unfavourable intermediate risk (NCCN) group with a visible dominant intraprostatic lesion (DIL), local dose escalation per DIL to 30 Gy will be performed.
  Interventions: Radiation: Single Dose Radiotherapy

INTERVENTIONS:
Radiation: Single Dose Radiotherapy — Procedure: external-beam radiotherapy (EBRT) on a linear accelerator with a dose 24 Gy in one session using technique of image-guided volumetric intensity modulation arc therapy (VMAT-IGRT) and a set of dedicated devices that ensure target immobilization and reproducibility of prostate anatomical localization during treatment. A special air-filled endorectal balloon will be used for immobilization of the prostate and anatomical reproducibility of organs at risk during treatment. A Foley catheter will be used to ensure reproducibility of the urethral position and online tracking of the prostate gland position during treatment. A special external immobilization system, including patient positioning on a patient transfer trolley, which allows for patient transfer without removing the endorectal balloon and urinary catheter from the table at all stages of pre-radiation preparation (MR, CT, Positron emission tomography (PET) / CT simulation) and during the treatment.

SUMMARY:
The goal of this study is to assess the feasibility of high-dose radiotherapy (Single-Dose Radiotherapy, SDRT) of 24 Gy in patients with localized low and intermediate risk prostate cancer using a special system of internal and external immobilization of the prostate gland.

Patients eligible for this study are classified according to the National Comprehensive Cancer Network (NCCN) guidelines as low or intermediate risk prostate cancer (Stage T1-T2c and/or Prostate Specific Antigen (PSA) level ≤20 ng/mL and/or Gleason score of ≤7).

The study will examine the technical feasibility of image-guided volumetrically-modulated arc therapy (VMAT-IGRT) with an emphasis on normal tissue sparing and precision of radiation delivery using dedicated devices (an air-filled endorectal balloon and a Foley catheter) that ensure target immobilization and reproducibility of prostate anatomical localization using a special external patient immobilization system, including patient placement on the patient transfer trolley, which allows patient transfer without removing the endorectal balloon and urinary catheter during all stages of simulation and treatment planning (MR, CT, Positron emission tomography (PET) / CT-simulation) and during the treatment session on the linear accelerator.

Previously untreated patients with localized prostate cancer of the low risk and favorable intermediate risk (NCCN) groups will receive SDRT at a dose of 24 Gy. In patients from the unfavourable intermediate risk (NCCN) group with a visible dominant intraprostatic lesion (DIL), local escalation of the DIL dose to 30 Gy will be performed.

Patients will be followed up at one week and one month after completion of treatment, then every 3 months for 24 months (+/- 4 weeks), and every 6 months thereafter. Evaluation of early and late adverse events will focus, although not exclusively, on the genitourinary and gastrointestinal toxicity, primarily the rectal toxicity. Serum prostate-specific antigen (PSA) levels will be determined according to the clinical follow-up schedule. Multiparametric magnetic resonance imaging (mpMRI) with intravenous contrast will be performed at baseline and at 6-, 12-, and 24-months post-intervention. Participants of the study will be followed up for at least 2 years after treatment.

DETAILED DESCRIPTION:
This study evaluates the clinical outcomes and potential adverse events associated with external beam single-dose radiotherapy (SDRT) using a dedicated internal and external target immobilization system in patients with low- and intermediate-risk localized prostate adenocarcinoma.

The findings from recently published randomized trial demonstrate that five-fraction SBRT is a robust and viable alternative to moderately fractionated radiotherapy for prostate cancer, demonstrating equivalent efficacy with enhanced convenience for patients. The high 5-year biochemical control rates, tolerability of treatment, coupled with the significant advancements in radiotherapy delivery, underscore the potential of Stereotactic Body Radiation Therapy (SBRT) use in prostate cancer treatment.

The feasibility of Single-Dose RadioTherapy (SDRT) in localized prostate cancer was tested in the randomized PROSINT trial comparing 5-session ultra-hypofractionated radiotherapy course with a Single Dose of 24 Gy radiotherapy. The 4-year results of this trial were recently published. The adverse event profile in both comparison groups was exceptionally good, with no severe adverse events of 3 or higher according to the NCI CTCAE v.4.0 scale and similar biochemical tumor response to both treatment regimens.

Patients enrolled in this trial will undergo volumetric intensity modulation arc therapy (VMAT-IGRT) using state-of-the-art dosimetric radiation therapy planning and quality assurance procedures with an emphasis on normal tissue sparing and precision of radiation delivery using dedicated devices that ensure target immobilization and reproducibility of prostate anatomical localization. A special endorectal balloon filled with air will be used for immobilization of the target in the prostate gland and anatomical reproducibility, while a urethral Foley catheter will be used to ensure reproducibility of the urethral position and online tracking of the prostate gland position (during the entire radiotherapy session). The study will also examine the technical feasibility of using a special external patient immobilization system, including patient positioning on a patient transfer trolley, which allows for patient transfer without removing the endorectal balloon and urinary catheter from the table at all stages of pre-radiation preparation (MR, CT, Positron emission tomography (PET) / CT simulation) and during the treatment session on the linear accelerator. Previously untreated patients with localized prostate cancer in the low risk and favorable intermediate risk (NCCN) groups will receive SDRT at a dose of 24 Gy. In patients in the unfavourable intermediate risk (NCCN) group with a visible dominant intraprostatic lesion (DIL), local dose escalation per DIL to 30 Gy will be performed.

Patients will be followed up at one week and one month after completion of treatment, then every 3 months for 24 months (+/- 4 weeks), and every 6 months thereafter. Evaluation of early and late adverse events will focus, although not exclusively, on the genitourinary and gastrointestinal tracts, primarily the rectum. Serum prostate-specific antigen (PSA) levels will be determined according to the clinical follow-up schedule. Multiparametric magnetic resonance imaging (mpMRI) with intravenous contrast will be performed at baseline and at 6-, 12-, and 24-months post-intervention. The study participants will be followed up for at least 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Signed study specific informed consent form;
* Histologic confirmation of adenocarcinoma of the prostate by biopsy;
* Biopsy Gleason score ≤ 7;
* Up to 6 months of previous hormonal therapy is allowed (but not required);
* PSA ≤ 20 prior to hormone therapy (if given);
* No direct evidence of regional or distant metastases after appropriate staging studies (CT, MRI, 68Ga-Prostate-Specific Membrane Antigen (PSMA) Positron emission tomography (PET) / CT)
* Age ≥ 18;
* Performance Status 0-2;
* International Prostate Symptom Score (IPSS) must be ≤ 15 (alpha blockers allowed)
* Computerized Tomography (CT) or Magnetic Resonance Imaging (MRI) or Ultrasound-based volume estimation of prostate gland ≤ 100 cc

Exclusion Criteria:

* Positive lymph nodes or metastatic disease from prostate cancer on imaging studies (CT, MRI, 68Ga-Prostate-Specific Membrane Antigen (PSMA) Positron emission tomography (PET) / CT);
* Tumour Clinical stage T3 or T4 on MRI;
* Gleason score > 7;
* PSA > 20 ng/mL;
* Previous pelvic radiotherapy;
* Previous surgery for prostate cancer;
* Recent transurethral resection of the prostate (TURP) (less than 3 months);
* Previous hormonal therapy given for more than 6 months prior to therapy;
* Prior invasive malignancy unless disease free for a minimum of 3 years;
* Previous significant urinary obstructive symptoms;
* Significant psychiatric illness;
* Ultrasound or CT or MRI estimate of prostate volume > 100 cc;
* Severe, active co-morbidity.
* Inability to fulfill all dosimetric criteria for target dose coverage and restrictions for the organs at risk according to study protocol;

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2024-07-24 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Number of patients with treatment-related adverse events as assessed by Common Toxicity Criteria for Adverse Effects v4.0 | 2 years
  Assessment of treatment related adverse events as measured by Common Toxicity Criteria for Adverse Effects v4.0 over a 5 year time frame.
Concentration of serum PSA | 2 years
  Changes of serum PSA after treatment
Biochemical relapse-free survival (bRFS) | 2 years
  Biochemical relapse-free survival rate (Phoenix Definition)

SECONDARY OUTCOMES:
Expanded Prostate Cancer Index Composite (EPIC) Questionnaire to measure quality of life | 2 years
  Quality of life is measured on a scale of 0 to 100, with higher scores representing a higher quality of life.
International Index of Erectile Function (IIEF) Questionnaire to assess sexual function | 2 years
  Sexual function is measured on a scale of 0 to 75, with higher scores representing higher sexual function.
Primary prostate tumor response based on multi-parametric MRI imaging | 2 years
  Assessment of tumor response based on prostate multi-parametric MRI changes after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Sergey Usychkin, MD, Principal Investigator — Chief Radiation Oncologist
Locations (1):
- The Branch of Hadassah Medical LTD, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No